CLINICAL TRIAL: NCT02169609
Title: Phase II Single Arm Study to Assess Dinutuximab (Ch 14.18) Combined With the Cytokines Granulocyte-macrophage Colony Stimulating Factor (GM-CSF) and IL-2 in Patients With High-risk Neuroblastoma Not Eligible to Other Immunotherapy Trials
Brief Title: Safety Study of Dinutuximab Combined With Immunotherapy to Treat Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSJD-HR-NB-Ch14.18
Record Dates: First submitted 2014-06-12; First posted 2014-06-23 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Neuroblastoma; Neoplasm, Residual; Effects of Immunotherapy
Keywords: Neuroblastoma; Immunotherapy; Dinutuximab
MeSH Terms: conditions — Neuroblastoma; Neoplasm, Residual | interventions — dinutuximab; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Isotretinoin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dinutuximab. Immunotherapy (Experimental): Dinutuximab will be administered at 17.5 mg/m2/day for 4 days up to 5 courses. Each dose should be infused IV over approximately 10 hours.
  Immunotherapy (sargramostim + isotretinoin + interleukin2) Sargramostim will be administered at 250 micrograms/m2/d by subcutaneous (SC) injection daily from Day 0 through 13 (daily with the infusion of Dinutuximab and for 3 days before and 7 days afterward).
  Isotretinoin (13-cis-retinoic acid, or RA) (160mg/m2/day or 5.33mg/kg/day if < 12kg) PO divided into 2 doses daily x 14 days.
  Interleukin-2 (IL-2) 3 MIU/m2/day will be given by continuous infusion for 4 days during the first week of each course 2 and 4 given on Days 0 - 3
  Interventions: Drug: Dinutuximab. Immunotherapy

INTERVENTIONS:
Drug: Dinutuximab. Immunotherapy — Patients will receive 5 courses of Dinutuximab + GM-CSF + IL2 at intervals of 28 days for all courses. In addition, all patients will receive isotretinoin (13-cis-retinoic acid, or RA) at 160 mg/m2/dose twice a day for 14 days every 28 days, for 6 courses.
  Patients come off study if progressive disease develops at any time after cycle 1 or life-threatening grade 4 toxicity occurs clearly attributable to Immunotherapy.
  Other Names: Ch14.18; Sargramostim; GM-CSF; Isotretinoin; 13-cis-retinoic acid, or RA; Interleukin-2 (IL-2)

SUMMARY:
The purpose of this study is to evaluate safety of the triple COG schema with the monoclonal antibody Dinutuximab + cytokines (GM-CSF and IL2) and isotretinoin (13-cis-retinoic acid, or RA) in patients with high-risk neuroblastoma.

DETAILED DESCRIPTION:
Assess toxicity and safety of subcutaneous GM-CSF and iv IL-2 in enhancing Dinutuximab-mediated ablation of Bone Marrow (BM) disease in patients with high-risk neuroblastoma who have achieved a Complete Response or Very Good Partial Response of the macroscopic disease in the investigators institution.

Assess response of minimal residual disease (MRD) of the anti-GD2 monoclonal antibody Dinutuximab combined with granulocyte-macrophage colony stimulating factor (GM-CSF) and IL-2 in patients with high-risk neuroblastoma (NB). More precisely, to apply real-time quantitative RT-PCR to test the hypothesis that minimal residual disease content of BM after the first treatments with dinutuximab/GM-CSF has significant prognostic impact on relapse-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of neuroblastoma as defined by international criteria by histopathology or bone marrow metastases. Patients age must be less than 18 years at the time of initial diagnosis.
2. Neuroblastoma, as defined by risk-related treatment guidelines and the International Neuroblastoma Staging System, stage 4 with (any age) or without (>18 months) MYCN-amplification, or MYCN-amplified neuroblastoma other than stage 1, or high-risk neuroblastoma defined based on the 3-gene molecular profile developed at our institution (Garcia I, et al. CCR 2012).

   * Group 1 patients have neuroblastoma (as defined above) resistant to standard therapy, as evidenced by incomplete response in bone marrow, but no MIBG-avid soft tissue or bone tumor and no progressive disease.
   * Group 2 patients have no evidence of measurable disease

     3 - Patients must have a Lansky or Karnofsky Performance Scale score of > 50% and patients must have a life expectancy of > 2 months.

4- Pre-enrollment tumor survey: Prior to enrollment a determination of residual disease must be Performed (Tumor imaging studies including CT or MRI, MIBG scan, bone marrow aspiration & biopsy, and blood and bone marrow samples). This disease assessment is required for eligibility.

5 - Patients must have adequate organ functions at the time of registration:

* Hematological: Total absolute phagocyte count (APC = neutrophils + monocytes) is at least 1000/microL
* Renal: Adequate Renal Function Defined As: Creatinine clearance or radioisotope GFR > 70 mL/min/1.73 m2 or serum creatinine based on age/gender.
* Hepatic- total bilirubin < 1.5 x normal, and SGPT (ALT) < 5 x normal. Veno-occlusive disease, if present, should be stable or improving.
* Cardiac- shortening fraction of > 30% by echocardiogram, or if shortening fraction abnormal, ejection fraction of > 55% by gated radionuclide study.
* Pulmonary- FEV1 and FVC > 60% of predicted by pulmonary function test. For children who are unable to do PFTs, no evidence of dyspnea at rest, no exercise intolerance.
* Central nervous system- Patients with seizure disorder may be enrolled if on anticonvulsants and wellcontrolled. CNS toxicity < Grade 2.

  6 - Females of childbearing potential must have a negative pregnancy test. Patients of childbearing potential must agree to use an effective birth control method. Female patients who are lactating must agree to stop breast-feeding.

  7 - Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

1. - Existing severe major organ dysfunction, i.e., renal., cardiac, hepatic, neurologic, pulmonary, or gastrointestinal toxicity ≥ grade 3.
2. - Progressive disease or MIBG-avid soft tissue/bone tumor.
3. - Active life-threatening infection.
4. - Inability to comply with protocol requirements.
5. - Patient is eligible for SIOP HR-NB-01 protocol (= newly diagnosed high-risk neuroblastoma patient in a center where the SIOP protocol is open for enrollment).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2016-12-26 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Expected, 7 months from treatment initiation. From IC signature, every day during immunotherapy treatment (Cycles 1 to 5), day 1 of cycle 6. From patient consent signature up to 30 days after administration of the last dose of study drug.
  Type, incidence, severity, timing, seriousness, and relatedness; of reported AEs, physical examinations, and laboratory tests. Toxicity will be graded and tabulated by the NCI-CTCAE v 4.0.

SECONDARY OUTCOMES:
Relapse-free survival | Anticipated, 2 years from study treatment initiation. From IC signature, every 3 months, up to 2 years (anticipated).
  Rate of BM response for patients with detectable minimal residual disease in the BM after the first treatments with Dinutuximab/GM-CSF and relation with relapse-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Mora, MD, Principal Investigator — Hospital Sant Joan de Deu, Barcelona
Locations (1):
- Hospital Sant Joan de Deu, Barcelona, Spain